CLINICAL TRIAL: NCT00291564
Title: Ensure Cardiac Resynchronization Therapy Study
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Other Study IDs: 239
Record Dates: First submitted 2006-02-10; First posted 2006-02-14 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Heart Failure
Keywords: Observational; Heart Failure; Continuous Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy Devices

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy Device

SUMMARY:
The purpose of this study is to gather information on how doctors program particular settings on cardiac resynchronization therapy implantable cardiac defibrillators (CRT-Ds), to analyze how these settings affect the amount of cardiac resynchronization therapy (CRT) patients receive and to evaluate the therapy approach for converting abnormally fast heartbeats into normal heartbeats. There are no experimental devices or procedures involved in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is indicated for a Medtronic CRT-D system
* Patient is willing to sign Permission for Access to and Use of Health Information form
* Patient is willing and able to comply with follow-up visits through six months

Exclusion Criteria:

* Patient has a life expectancy of less than 6 months
* Patient is participating in any concurrent study that could confound the results for either study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430
Dates: Start 2004-05; Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Thompson, MD, Principal Investigator — Tennessee Cardiovascular Research Institute
Locations (32):
- United States (32):
  - Birmingham, Alabama
  - Newport Beach, California
  - Trumbull, Connecticut
  - Daytona Beach, Florida
  - Augusta, Georgia
  - Kankakee, Illinois
  - Indianapolis, Indiana
  - Des Moines, Iowa
  - Owensboro, Kentucky
  - New Orleans, Louisiana
  - Salisbury, Maryland
  - Burlington, Massachusetts
  - Detroit, Michigan
  - Traverse City, Michigan
  - Minneapolis, Minnesota
  - Mexico, Missouri
  - Omaha, Nebraska
  - Bridgewater, New Jersey
  - Englewood, New Jersey
  - Charlotte, North Carolina
  - Dayton, Ohio
  - Lyndhurst, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Abington, Pennsylvania
  - Doylestown, Pennsylvania
  - Columbia, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - Fairfax, Virginia
  - Richmond, Virginia
  - Seattle, Washington